CLINICAL TRIAL: NCT06792123
Title: The Effect of Virtual Reality Application Applied to Patients with Total Knee Replacement At Different Times on Anxiety and Recovery Quality
Brief Title: Effect of Virtual Reality Application Applied to Patients with Total Knee Replacement At Different Times
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Özge İşeri (Other)
Responsible Party: Sponsor-Investigator, Özge İşeri, Assistant Professor, Ondokuz Mayıs University, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMUKAEK 2023/423; Ondokuz Mayıs University (Other: Ondokuz Mayıs University)
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Recovery Quality
Keywords: virtual reality; anxiety; recovery quality; total knee replacement; nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1 (Experimental): pre-op VR application group
  Interventions: Other: pre-op VR application group
- Group 2 (Experimental): Intra-op VR application group
  Interventions: Other: intra-op VR application group
- Control (No Intervention): Standart care and treatment

INTERVENTIONS:
Other: pre-op VR application group — VR application group during preoperative process
  Arms: group 1
Other: intra-op VR application group — VR application group during intraoperative process
  Arms: Group 2

SUMMARY:
The aim of this study was to examine the effect of virtual reality application on anxiety and quality of recovery at different times (preoperatively and intraoperatively) in patients undergoing total knee replacement.

DETAILED DESCRIPTION:
The elderly population in the world and in our country is gradually increasing and the aging process is prolonged due to the prolongation of life expectancy. Osteoarthritis is one of the important obstacles limiting low quality of life and physical freedom in this aging process. It is estimated that osteoarthritis affects over 250 million people worldwide. Osteoarthritis is one of the important causes of severe pain and disability due to limitation of mobility, and this disease is a disease that causes deterioration in the psychological well-being of individuals and a low quality of life. The presence of symptoms characterized by joint pain, stiffness and limitation of movement in osteoarthritis negatively affects the quality of life of individuals. One of the most common problems in our country is osteoarthritis of the knee. In the treatment of osteoarthritis of the knee, total knee replacement surgery is performed as a last resort if pharmacologic and non-pharmacologic methods do not yield a positive response. Patients with total knee replacement may be exposed to anxiety and pain in this process. In previous studies, positive results were found when the effects of virtual reality application on pain were examined. The aim of this study was to examine the effect of virtual reality application on anxiety and quality of recovery at different times (preoperatively and intraoperatively) in patients undergoing total knee replacement. In previous studies, it was determined that virtual reality application was mostly applied preoperatively and examined pain and vital signs. There are no studies on quality of recovery

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* No psychiatric medication
* No mental and cognitive disabilities
* Those who underwent Total Knee Replacement,

Exclusion Criteria:

* Patients with visual and hearing impairment
* Receiving general anesthesia
* Experiencing complications during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Pre-test before surgery; post-test two hours after surgery
  Beck Anxiety Scale
Recovery quality | Pre-test before surgery; post-test two hours after surgery
  quality of recovery-15 (QoR-15)

CONTACTS AND LOCATIONS:
Overall Officials: Özge İşeri Assistant Professor, PhD, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs Unıversity, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Since this is a master thesis, the results will be shared at the end of the thesis